CLINICAL TRIAL: NCT04220112
Title: Comparing Real-time fMRI Neurofeedback Versus Sham for Altering Limbic and Eating Disturbances in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PSYCH-2019-28137
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Anorexia; Anorexia Nervosa
MeSH Terms: conditions — Anorexia; Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Time Functional MRI (rt-fMRI) (Experimental): Real-time fMRI (rt-fMRI) neurofeedback (focused on amygdala down-regulation) intervention
  Interventions: Procedure: Real-Time Functional Magnetic Resonance Imaging (RT-fMRI)
- Sham (Sham Comparator): Sham-controlled group
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Procedure: Real-Time Functional Magnetic Resonance Imaging (RT-fMRI) — RT-fMRI neurofeedback targeting down-regulation of the amygdala
  Arms: Real Time Functional MRI (rt-fMRI)
Procedure: Sham Procedure — RT-fMRI with feedback non-contingently tied to their activation patterns (activation patterns from a prior participant)
  Arms: Sham

SUMMARY:
The goal of the purposed research is to extend prior work (STUDY00003758: Real-time fMRI Neurofeedback to Alter Limbic Disturbances in Anorexia Nervosa) on real-time fMRI (rt-fMRI) neurofeedback (focused on amygdala down-regulation) as an innovative neurocircuitry-targeted intervention for anorexia nervosa (AN). This project will include randomization to rt-fMRI or a sham controlled group to answer the following important unresolved question: Does a patient-led procedure aimed at altering brain activity impact limbic circuit function and key eating disorder and psychiatric symptoms in AN above the effect of a matched, but non-targeted sham condition?

DETAILED DESCRIPTION:
Aim 1: Establish that rt-fMRI neurofeedback of limbic activity can correct neural disturbances in AN. Hypothesis 1: Compared to the sham group, the amygdala neurofeedback group will show reduced amygdala activation to aversive images, which will increase with repeated training. This effect will generalize to non-neurofeedback test runs. Hypothesis 2: Compared to the sham group, the amygdala neurofeedback group will exhibit enhanced task and resting amygdala-prefrontal cortex (PFC) connectivity, which will increase with repeated training. Enhanced amygdala-PFC connectivity will be associated with less amygdala reactivity to aversive images during the emotion regulation task.

Aim 2: Identify the impact of rt-fMRI neurofeedback targeting limbic functioning on symptoms of AN. Hypothesis 1: Compared to the sham group, the amygdala neurofeedback group will exhibit improvements in self-reported emotion regulation and eating disorder symptoms over the study visits. Hypothesis 2: Compared to the sham group, the amygdala neurofeedback group will engage in less restrictive eating (i.e., will consume more calories) at a post-training test meal. Hypothesis 3: Across groups, decreased aversive amygdala reactivity and enhanced amygdala-PFC connectivity will predict reduced emotion dysregulation and eating disorder symptoms, and less restriction.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of AN, with the exception of body image disturbance and intense fear of weight gain
* Ability to read and speak in English
* Right-handed

Exclusion Criteria:

* Medical instability or current pregnancy (self-reported)
* Acute suicidality, current substance use disorder, psychosis, or mania
* Contraindication for fMRI as determined by CMRR safety screening standards
* History of neurological disorder/injury (e.g., stroke; head injury with > 10 minutes loss of consciousness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Eating Disorder Symptoms Scale (CHEDS) | 2 months
  CHEDS is a 35-item self-report measure designed to assess eating disorder symptom changes over a short-term (i.e. weekly) time span. Items are presented using a Likert response format in which symptoms are rated from 0 (never) to 4 (always) during the past week. Total score is a sum of the 35 item scores.
Change in Body Mass Index (BMI) | 2 months
  Change in body mass index (BMI) from baseline to end (2 months). BMI is calculated as body weight (in kg) divided by height (in cm) squared. BMI is reported in kg/(cm^2).
Test Meal Caloric Intake | 2 months
  Caloric consumption (in kilocalories) from a laboratory test meal

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haynos, PhD, Principal Investigator — University of Minenesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No